CLINICAL TRIAL: NCT02325375
Title: Inflammation in Amyotrophic Lateral Sclerosis - a Study of Soluble Cluster of Differentiation 163 in the Cerebrospinal Fluid
Brief Title: sCD163 in ALS Patients
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: ALS CD163; 1-10-72-348-14 (Other: The National Committee on Health Research Ethics (Denmark))
Record Dates: First submitted 2014-12-16; First posted 2014-12-25 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2014-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; spinal fluid; CD163
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Spinal Puncture; Blood Specimen Collection

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — spinal fluid and blood sample for identification of different factors
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- ALS newly diagnosed
  Interventions: Procedure: lumbar puncture for spinal fluid and blood sample
- ALS treated
  Interventions: Procedure: lumbar puncture for spinal fluid and blood sample
- controls
  Interventions: Procedure: lumbar puncture for spinal fluid and blood sample

INTERVENTIONS:
Procedure: lumbar puncture for spinal fluid and blood sample — lumbar puncture for spinal fluid and blood sample

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a fatal disease with progressive muscle weakness leading to severe disability and eventually death.Since the diagnosis relies on clinical features and electromyographic abnormalities, which may occur rather late in the disease course, there is a need to identify diagnostic tests that can confirm or exclude the diagnosis of ALS in the earlier phase of the disease.

More recently, there are studies suggesting neuroinflammation to play a role for the development of ALS. Cluster of differentiation 163 is found to be up regulated in a large range of inflammatory diseases.

At the investigators lab, pilot data (Kallestrup M et al, unpublished data) has shown promising results. There was an increased level of cluster of differentiation 163 (sCD163) in cerebrospinal fluid in 7 patients with ALS compared with controls.

The purpose of the investigators study is to define the concentration of sCD163 in the cerebrospinal fluid and serum in patients with ALS compared with controls (patients with unspecified neurological symptoms). Furthermore, the investigators will define the concentrations of protein, glucose, immunoglobulin G index and other factors in the spinal fluid.

DETAILED DESCRIPTION:
Introduction Amyotrophic lateral sclerosis (ALS) is a fatal disease with progressive muscle weakness leading to severe disability and eventually death. It is the most common form of motor neuron diseases and involves both the upper and lower motor neurons. The median survival from debut of symptoms to dead is approximately 3 years.

Since the diagnosis relies on clinical features and electromyographic abnormalities, which may occur rather late in the disease course, there is a need to identify diagnostic tests that can confirm or exclude the diagnosis of ALS in the earlier phase of the disease.

ALS is a neurodegenerative disease, however the pathogenesis is not well established. The causes are probably multifactorial and a complex interaction between genetic factors and dysfunction of vital molecular pathways concerning the dominantly inherited c9orf72 gene and impaired glutamate uptake in astrocytes (EAAT2-receptor) from the synaptic cleft and thereby glutamate excitotoxicity. This glutamate excitotoxicity may cause oxidative stress, voltage-gated persistent sodium channels and activation of microglia resulting in secretion of proinflammatory cytokines.

More recently, there are studies suggesting neuroinflammation to play a role for the development of ALS. A study from 2012 (a mouse model of ALS, that overexpress mutant superoxide dismutase (mSOD1)), has documented that microglia can both protect and injure the motor neurones depending on which phenotype of the microglia is activated. It seems like it is a continuum between the protective M2 phenotypic state (disease onset) and the neurotoxic M1 phenotypic state (disease end-stage). Furthermore, at disease onset the mice expressed higher levels of Ym1, CD163 and brain-derived neurotrophic factor (markers of M2).

Of other molecular mechanisms, it is worth to mention the structural and functional abnormalities of mitochondria, impairment of axonal transport systems and endosomal trafficking and induction of the endoplasmic reticulum stress response although they appear to be secondary events in ALS. The net result is degeneration of motor neurones in cerebral cortex, the cranial nerve nuclei, the anterior horn of the spinal cord and the corticospinal tracts. The only present treatment available is Riluzole that has proven to extend life or time to onset of serious respiratory problems in patients with ALS. The mode of action for Riluzole still has to be determined, possibly the dynamic is an inhibition of glutamate release from the presynaptic neuron. (1,2,3,4,5,6) Though it seems that the inflammatory process is a secondary event, it seems to be critical for neuronal degeneration. In a study, ALS pathology was sought to be reduced through central nervous system targeted glucocorticoid and succeeded by reducing brainstem pathology in mouse models of ALS. Of different biomarkers, inflammatory markers have also been tested: the interleukin-1 family cytokines. Among them only total interleukin-18, its endogenous inhibitor interleukin-18BP, and the active form of the cytokine (free interleukin-18) were significantly higher in the ALS patients than in controls. The cytokine showed no correlation to the different clinical forms of ALS or the clinical setting of the disease. Cytokines have also been tried as neuroprotective agents. Erythropoietin (EPO) is known as the growth factor that maintains the number of circulating erythrocytes. However, the biological role of EPO has been expanded to other cells, such as neurons, microglia, and astrocytes in the brain. EPO seems to suppress the proinﬂammatory cytokines during disease progression, maintain the anti-inﬂammatory cytokines until the late symptomatic stage and finally seems to delay symptom onset and preserve number of motor neurons. (7,8,9,10) Cluster of differentiation 163 (CD-163) - a new way to monitor inflammation in ALS? CD-163 is a scavenger receptor (recognizes and uptakes macromolecules) which marks the monocyte-macrophage activation. CD163 works for macrophages as a receptor for hemoglobin-haptoglobin complexes. The soluble form of the receptor is called sCD163 and is found in plasma and cerebrospinal fluid, where it is found to be up regulated in a large range of inflammatory diseases.

Strongly increased values (>20mg/l) is seen in diseases like macrophage activating syndrome,hemophagocytic syndrome and acute hepatic failure. Furthermore, the level of sCD163 reflects the activity of the disease. Patients with increasing and high values are found to have unfavorable prognosis. Increased values (5-20 mg/l) are seen in hepatic disease, sepsis and Gaucher's disease. Septic patients with values greater than 10 mg/l have a 10 times greater risk of fatal outcome. Values which is increased a little (3-5 mg/l) is often seen in inflammatory of infectious conditions and in cancer. (11,12,13,14) Pilot data At the investigators lab, pilot data (Kallestrup M et al, unpublished data (15)) has shown promising results. There was an increased level of sCD163 in cerebrospinal fluid in 7 patients with ALS compared with controls. Furthermore, both definite and probable ALS patients have an increased level of sCD163. These results suggest a larger study to be performed evaluating patients with ALS at early as well as later stages of the disease.

Hypothesis Patients with ALS have up-regulated levels of sCD-163 in their cerebrospinal fluid and serum compared with healthy subjects and the level is related to the severity of the disease.

Purpose To define the concentration of sCD-163 in the cerebrospinal fluid and serum in patients with ALS compared with controls (patients with unspecified neurological symptoms). Furthermore, we will define the concentrations of protein, glucose, immunoglobulin G index and other factors in the spinal fluid.

Method Study population The study population will be all patients with established and suspected ALS at the Department of Neurology, Aarhus University Hospital.

Patients with established ALS who participate will undergo lumbar puncture as a part of this study. Subjects suspected to suffer from ALS will undergo lumbar puncture as a part of their diagnostic work up and the level of sCD163 in their cerebrospinal fluid will be analysed.

At the Department of Neurology, Aarhus University Hospital there are approximately 80 patients with established ALS. We expect that 50 of these patients are willing to participate and are eligible for inclusion (31-08-2015). Furthermore, we expect to include 8 patients who will be diagnosed with ALS at Department of Neurology, Aarhus University Hospital during the study period.

The controls include patients with various neurological symptoms or diseases who will undergo a lumbar puncture at the Department of Neurology at Aarhus University Hospital as part of their diagnostic work-up irrespective of this study. In the final analyses only controls will be included who end up having either no neurological disease or a neurological disease which is believed not to involve the spinal fluid. We expect to include 40-50 controls.

Recruitment Participants will receive written and oral information about the study. The oral information will take place at Department of Neurology, Aarhus University Hospital. Moreover, the pamphlet "Forsøgspersoners rettigheder i et sundhedsvidenskabeligt forskningsprojekt" will be handed out. Consultants at the department of neurology will give the information, to patients with suspected ALS. Controls and patients with established ALS will receive information from the doctors at the department of Neurology and research year student Anne Sofie Vinther.

It is possible to bring a companion and the participants are offered at least 24 hours to consider participation.

Access to patient records will be requested, which will be provided in the written information material.

If new knowledge about disadvantages of participating in the study appears the participants will be informed immediately. Moreover, the participant will be informed if evaluations during the study bring knowledge about the general health status of the patient, unless this has been clearly rejected by the patient.

By the end of the study it is possible for participants to contact the study coordinator to get information about study results.

All participants will receive information about the research project and will be asked to give their content to participation. The participation implies extraction of 5-6 ml spinal fluid and a blood sample (30ml), which will be used for analysis of sCD-163.

Participants will not receive any form of payment, but can receive compensation for transportation.

Inclusion criteria:

ALS Patients diagnosed with ALS and patients suspected to have ALS. Age >18 Controls Age >18

Exclusion criteria (for all groups):

Acute infections including neuroinfection Other disorders known to have elevated levels of sCD163 Disorders or treatments that contraindicate a lumbar puncture. Other established neurological disorders. At all times during the diagnostic work-up and consequently in the research project we will do this with respect for the patients mental and physical condition. The research project will be carried out according to the Act on Processing of Personal Data and, furthermore, the project will be submitted to the common regional information system for Region Midtjylland.

Analysis The spinal fluid and the serum will be analysed at the Department of Clinical Biochemistry, Aarhus University Hospital. The spinal fluid and blood samples will be deposited in a research biobank at Aarhus University Hospital. It is planned that all biochemical analyses will be performed when all samples are collected. At the end of the project, the samples will be pseudo anonymised. Due to the possibility of developing new knowledge in this area, the samples will be deposited in the biobank 5 years after this project has been finished.

The concentrations of sCD-163 in spinal fluid and serum will be analyzed by already established techniques at the Department of Clinical Biochemistry, Aarhus University Hospital.

Examination The examination consists of a medical history and a clinical examination. We use the Revised ALS functional rating scale (ALSFRS-R), which is at rating instrument for monitoring the progression of disability in patients with ALS. Information from the medical record will be included and used in this project including past medical history, actual use of drugs, results of biochemical analyses and brain imaging, results from the ALSFRS-R, results from the electromyography, abnormalities at the clinical examinations and the conclusions from the diagnostic work-up.

Power and Statistical analyses Since the investigators pilot data (n=7) showed a 50% increase in the level of CD163 in the cerebrospinal fluid in ALS patients inclusion of 40 patients is expected to enable detection of smaller difference also in serum and relations between CD163 and clinical findings.

The program ANOVA will be used for statistical analyses. Parametric or non-parametric tests will be used depending of the normal distribution of data. In all statistical analysis a 5% level of significance will be used.

Perspectives It is of importance to identify prognostic biomarkers in ALS. The pathology of ALS is still unknown but it seems that inflammation is a crucial factor in the process. In several studies, sCD163 has shown to be up regulated in a large range of inflammatory diseases and together with the investigators promising pilot data sCD163 is a potential marker for ALS. (4) The assessment of drug efficacy in ALS remains clinically based, relying on measuring the rate of disease progression through the utilization of the ALS rating scale-revised (ALSFRS-R). Such clinical scales may be insensitive, especially in the early stages of the disease process. The development of reliable quantifiable biomarkers remains elusive in ALS, and development of prognostic biomarkers would be crucial for effective evaluation of a therapeutic agent in the early stages of development.

Ethical consideration The tests performed on the patients involved in this research project are lumbar puncture and blood samples.

It involves some risks to perform a lumbar puncture, which include post lumbar puncture headache with an incidence of 12 %, most common in younger patients. Most frequently, the headache has a short duration and it may be cured with application of a blood-patch. Moreover, lumbar puncture can cause temporary lumbar pain and an accumulation of blood underneath the skin. There is a very low risk of bleeding in the epidural space with compression of spinal nerves and an even lower risk of infections (meningitis or meningoencephalitis). However, it is important to underscore that lumbar puncture is part of routine diagnostic workup at the Department of Neurology at Aarhus University Hospital.

In consideration of the low risk involved in this project, the bad prognosis for the disease and the potential to improve diagnosis and treatment for future patients with ALS we consider this project to be ethically acceptable.

Publication Positive, negative as well as inconclusive results from this study will be published. The results will be written in an article for publication in an English written peer reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

* ALS and controls(lumbar puncture at our department)

Exclusion Criteria:

* <18 years
* Other CNS disease

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ALS, treated or newly diagnosed
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Concentrations of sCD-163 in patients with ALS. | day 1
Concentration of sCD163 in newly diagnosed compared with established ALS | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Vucic S, Rothstein JD, Kiernan MC. Advances in treating amyotrophic lateral sclerosis: insights from pathophysiological studies. Trends Neurosci. 2014 Aug;37(8):433-42. doi: 10.1016/j.tins.2014.05.006. Epub 2014 Jun 11. PMID 24927875
- [Background] Menon P, Kiernan MC, Vucic S. Biomarkers and future targets for development in amyotrophic lateral sclerosis. Curr Med Chem. 2014;21(31):3535-50. doi: 10.2174/0929867321666140601161148. PMID 24934359
- [Background] Liao B, Zhao W, Beers DR, Henkel JS, Appel SH. Transformation from a neuroprotective to a neurotoxic microglial phenotype in a mouse model of ALS. Exp Neurol. 2012 Sep;237(1):147-52. doi: 10.1016/j.expneurol.2012.06.011. Epub 2012 Jun 23. PMID 22735487
- [Background] Evans MC, Gaillard PJ, de Boer M, Appeldoorn C, Dorland R, Sibson NR, Turner MR, Anthony DC, Stolp HB. CNS-targeted glucocorticoid reduces pathology in mouse model of amyotrophic lateral sclerosis. Acta Neuropathol Commun. 2014 Jun 13;2:66. doi: 10.1186/2051-5960-2-66. PMID 24923195
- [Background] Italiani P, Carlesi C, Giungato P, Puxeddu I, Borroni B, Bossu P, Migliorini P, Siciliano G, Boraschi D. Evaluating the levels of interleukin-1 family cytokines in sporadic amyotrophic lateral sclerosis. J Neuroinflammation. 2014 May 23;11:94. doi: 10.1186/1742-2094-11-94. PMID 24884937
- [Background] Dumont AO, Goursaud S, Desmet N, Hermans E. Differential regulation of glutamate transporter subtypes by pro-inflammatory cytokine TNF-alpha in cortical astrocytes from a rat model of amyotrophic lateral sclerosis. PLoS One. 2014 May 16;9(5):e97649. doi: 10.1371/journal.pone.0097649. eCollection 2014. PMID 24836816
- [Background] Noh MY, Cho KA, Kim H, Kim SM, Kim SH. Erythropoietin modulates the immune-inflammatory response of a SOD1(G93A) transgenic mouse model of amyotrophic lateral sclerosis (ALS). Neurosci Lett. 2014 Jun 27;574:53-8. doi: 10.1016/j.neulet.2014.05.001. Epub 2014 May 10. PMID 24820540
- [Background] Kjaergaard AG, Rodgaard-Hansen S, Dige A, Krog J, Moller HJ, Tonnesen E. Monocyte expression and soluble levels of the haemoglobin receptor (CD163/sCD163) and the mannose receptor (MR/sMR) in septic and critically ill non-septic ICU patients. PLoS One. 2014 Mar 17;9(3):e92331. doi: 10.1371/journal.pone.0092331. eCollection 2014. PMID 24637679
- [Background] Etzerodt A, Moestrup SK. CD163 and inflammation: biological, diagnostic, and therapeutic aspects. Antioxid Redox Signal. 2013 Jun 10;18(17):2352-63. doi: 10.1089/ars.2012.4834. Epub 2012 Oct 19. PMID 22900885
- [Background] Moller HJ. Soluble CD163. Scand J Clin Lab Invest. 2012 Feb;72(1):1-13. doi: 10.3109/00365513.2011.626868. Epub 2011 Nov 7. PMID 22060747
- See also: Up To Date — http://www.uptodate.com/contents/search?search=ALS&x=0&y=0
- See also: About medication — http://pro.medicin.dk/Medicin/Praeparater/7115